CLINICAL TRIAL: NCT00625495
Title: An Open, Randomised Two Way Crossover Study Comparing the Effects of 40mg of Esomeprazole Adminstered Orally and Intravenously as a 3 Minute Injection on Basal and Pentrigastrin-stimulated Acid Output in Subjects With Symptoms of Gastroesophageal Reflux Disease (GERD)
Brief Title: Study Comparing the Effects of Esomeprazole Adminstered Orally and Intravenously on Basal and Pentrigastrin-stimulated Acid Output in Subjects With Symptoms of Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind, MD - Nexium Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D9615C00013
Record Dates: First submitted 2008-02-20; First posted 2008-02-28 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal reflux disease; Nexium; Esomeprazole; Administration methods.
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): IV Nexium
  Interventions: Drug: Esomeprazole
- 2 (Experimental): Oral Nexium
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — 40mg Intravenous infusion over 3 minutes
  Other Names: Nexium
  Arms: 1
Drug: Esomeprazole — 40mg Oral
  Other Names: Nexium
  Arms: 2

SUMMARY:
The purpose of this study is to examine the effects of Nexium at a dose of 40mg administered orally compared to intravenously on the maximum acid output in subjects with symptoms of Gastroesophageal reflux disease (GERD).

ELIGIBILITY:
Inclusion Criteria:

* Heartburn on 2 out of the last 7 days prior to screening or a diagnosis of GERD (with or without a diagnosis of Erosive eosphagitis).
* Body Mass Index within the limits specified in the protocol

Exclusion Criteria:

* History of esophageal, duodenal or gastric surgery
* History of severe liver disease.
* Any other significant disease or pathology judged to be clinically significant by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-09; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
To compare the maximum acid output during pentagastrin stimulation after 10 days of Nexium dosing administered orally with 10 days dosing via intravenous administration. | Every 10 days

SECONDARY OUTCOMES:
To compare basal acid output at steady state and when switching between Oral and IV adminstration of Nexium. | Post Day 10
To compare maximum acid output when switching between Oral and IV adminstration of Nexium | Post Day 10
Safety assessment via adverse event recording | At each visit

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca